CLINICAL TRIAL: NCT05030948
Title: A Physical Activity Intervention to Promote Cognitive Health, Cardiovascular Health and Sleep in Older Latinos
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Gloria Adriana Perez, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 844561; 1R01AG070351-01 (NIH)
Record Dates: First submitted 2021-07-30; First posted 2021-09-01 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Older Latinos; Cardiovascular Health; Sleep Quality; Cognitive Function; Community Health Worker; Walking; Physical Activity
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tiempo Juntos Intervention (Experimental): If assigned to this group, participants will take part in weekly 1-hour group sessions twice a week for 3 months. The sessions will be with a trained Community Health Worker that will involve group (5-6 participants) moderate-intensity walking. They will take place at community partner sites during times when all participants can attend. In case of adverse weather, indoor locations are available through community partners. Walks will reflect participant goals and abilities, initially lasting 10 minutes, with 5-minute stretching "warm-up" and 5-minute "cool down" exercises, for a total of 20 minutes. Walk duration will increase by 5 minutes/week to at least 30 minutes with program content delivery time decreasing to accommodate increased walk times within the 1-hour session. Upon completing the 3 months of physical activity sessions, for the next 3 months, they will receive motivational "booster" sessions delivered every other week via phone calls/text messaging.
  Interventions: Behavioral: Tiempo Juntos Intervention
- Attention Control (No Intervention): If assigned to this group, participants will take part in 1-hour group (5-6 participants) sessions delivered twice a week for 3 months. The sessions will be with a trained Community Health Worker or qualified staff that will involve reviewing education topics in Spanish related to adult health. They will take place at community partner sites or remotely during times when all participants can attend. In case of adverse weather, indoor locations, or remote options will be available. Upon completing the 3 months of education sessions, for the next 3 months, they will receive educational "booster" sessions delivered every other week via phone calls/text messaging.

INTERVENTIONS:
Behavioral: Tiempo Juntos Intervention — If assigned to this group, participants will take part in weekly 1-hour group sessions twice a week for 3 months. The sessions will be with a trained Community Health Worker that will involve group (5-6 participants) moderate-intensity walking. Upon completing the 3 months of physical activity sessions, for the next 3 months, they will receive motivational "booster" sessions delivered every other week via phone calls/text messaging.
  Arms: Tiempo Juntos Intervention

SUMMARY:
This study is a randomized, single-blind, controlled trial that will test a multilevel intervention, Tiempo Juntos para la Salud, (Time Together for Health) designed to promote moderate-intensity physical activity; theoretically grounded mediators; and secondary outcomes of cardiovascular health, sleep and cognitive function. Participants will have 4 visits over a year long period. Data collection will occur at baseline, 3 months, 6 months, and 12 months among 216 Spanish language-dominant Latinos aged 55 and older with Mild Cognitive Impairment (MCI) [Montreal Cognitive Assessment (MoCA) score 23 to 26 for Latino populations].

ELIGIBILITY:
Inclusion Criteria:

* Can provide informed consent
* 55+ years
* Self-identify as Hispanic/Latino
* Spanish as primary language
* Willing to attend intervention / education sessions
* Access to phone/cell
* less than 150 min of activity / week (sedentary)
* Montreal Cognitive Assessment (MoCA) score (score ≥ 23 to 26 for Latino populations)

Exclusion Criteria:

* Cannot provide informed consent
* Mobility disability
* Musculoskeletal problem / co-morbidity (prevents moderate PA)

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Physical Activity Frequency at 3 months | 12 weeks
  Number of activity sessions
Change from Baseline Physical Activity Frequency at 6 months | 24 weeks
  Number of activity sessions
Change from Baseline Physical Activity Frequency at 12 months | 48 weeks
  Number of activity sessions
Change from Baseline Physical Activity Intensity at 3 months | 12 weeks
  Light, moderate, or vigorous (determined by counts per minute)
Change from Baseline Physical Activity Intensity at 6 months | 24 weeks
  Light, moderate, or vigorous (determined by counts per minute)
Change from Baseline Physical Activity Intensity at 12 months | 48 weeks
  Light, moderate, or vigorous (determined by counts per minute)
Change from Baseline Physical Activity Duration at 3 months | 12 weeks
  Total time spent in activity (hours and minutes)
Change from Baseline Physical Activity Duration at 6 months | 24 weeks
  Total time spent in activity (hours and minutes)
Change from Baseline Physical Activity Duration at 12 months | 48 weeks
  Total time spent in activity (hours and minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria A Perez, PhD, CRNP, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Nursing, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snowden M, Steinman L, Mochan K, Grodstein F, Prohaska TR, Thurman DJ, Brown DR, Laditka JN, Soares J, Zweiback DJ, Little D, Anderson LA. Effect of exercise on cognitive performance in community-dwelling older adults: review of intervention trials and recommendations for public health practice and research. J Am Geriatr Soc. 2011 Apr;59(4):704-16. doi: 10.1111/j.1532-5415.2011.03323.x. Epub 2011 Mar 25. PMID 21438861
- [Background] Coelho FG, Gobbi S, Andreatto CA, Corazza DI, Pedroso RV, Santos-Galduroz RF. Physical exercise modulates peripheral levels of brain-derived neurotrophic factor (BDNF): a systematic review of experimental studies in the elderly. Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):10-5. doi: 10.1016/j.archger.2012.06.003. Epub 2012 Jun 29. PMID 22749404
- [Background] Sink KM, Espeland MA, Castro CM, Church T, Cohen R, Dodson JA, Guralnik J, Hendrie HC, Jennings J, Katula J, Lopez OL, McDermott MM, Pahor M, Reid KF, Rushing J, Verghese J, Rapp S, Williamson JD; LIFE Study Investigators. Effect of a 24-Month Physical Activity Intervention vs Health Education on Cognitive Outcomes in Sedentary Older Adults: The LIFE Randomized Trial. JAMA. 2015 Aug 25;314(8):781-90. doi: 10.1001/jama.2015.9617. PMID 26305648
- [Background] Bherer L, Erickson KI, Liu-Ambrose T. A review of the effects of physical activity and exercise on cognitive and brain functions in older adults. J Aging Res. 2013;2013:657508. doi: 10.1155/2013/657508. Epub 2013 Sep 11. PMID 24102028
- [Background] Chin AL, Negash S, Hamilton R. Diversity and disparity in dementia: the impact of ethnoracial differences in Alzheimer disease. Alzheimer Dis Assoc Disord. 2011 Jul-Sep;25(3):187-95. doi: 10.1097/WAD.0b013e318211c6c9. PMID 21399486
- [Background] Committee PAGA. Physical activity guidelines advisory committee scientific report. Washington, DC: US Department of Health and Human Services. 2018.
- [Background] Gonzales A, Keller C. Mi familia viene primero (My family comes first): Physical activity issues in older Mexican American women. Southern Online Journal of Nursing Research. 2004;5(4):21.
- [Background] Melillo KD, Williamson E, Houde SC, Futrell M, Read CY, Campasano M. Perceptions of older Latino adults regarding physical fitness, physical activity, and exercise. J Gerontol Nurs. 2001 Sep;27(9):38-46. doi: 10.3928/0098-9134-20010901-08. PMID 11820555
- [Background] Marquez DX, Neighbors CJ, Bustamante EE. Leisure time and occupational physical activity among racial or ethnic minorities. Med Sci Sports Exerc. 2010 Jun;42(6):1086-93. doi: 10.1249/MSS.0b013e3181c5ec05. PMID 19997031
- [Background] King AC, Castro C, Wilcox S, Eyler AA, Sallis JF, Brownson RC. Personal and environmental factors associated with physical inactivity among different racial-ethnic groups of U.S. middle-aged and older-aged women. Health Psychol. 2000 Jul;19(4):354-64. doi: 10.1037//0278-6133.19.4.354. PMID 10907654
- [Background] Marquez DX, Aguinaga S, Campa J, Pinsker EC, Bustamante EE, Hernandez R. A Qualitative Exploration of Factors Associated With Walking and Physical Activity in Community-Dwelling Older Latino Adults. J Appl Gerontol. 2016 Jun;35(6):664-77. doi: 10.1177/0733464814533819. Epub 2014 May 15. PMID 24832017
- [Background] Fox AA, Thompson JL, Butterfield GE, Gylfadottir U, Moynihan S, Spiller G. Effects of diet and exercise on common cardiovascular disease risk factors in moderately obese older women. Am J Clin Nutr. 1996 Feb;63(2):225-33. doi: 10.1093/ajcn/63.2.225. PMID 8561064
- [Background] Winkleby MA, Feldman HA, Murray DM. Joint analysis of three U.S. community intervention trials for reduction of cardiovascular disease risk. J Clin Epidemiol. 1997 Jun;50(6):645-58. doi: 10.1016/s0895-4356(97)00020-6. PMID 9250263
- [Background] Taylor WC, Baranowski T, Young DR. Physical activity interventions in low-income, ethnic minority, and populations with disability. Am J Prev Med. 1998 Nov;15(4):334-43. doi: 10.1016/s0749-3797(98)00081-6. PMID 9838976
- [Background] Piedra LM, Andrade FCD, Hernandez R, Trejo L, Prohaska TR, Sarkisian CA. Let's walk! Age reattribution and physical activity among older Hispanic/Latino adults: results from the inverted exclamation markCaminemos! Randomized trial. BMC Public Health. 2018 Aug 3;18(1):964. doi: 10.1186/s12889-018-5850-6. PMID 30075709
- [Background] Perez A, Fleury J, Belyea M. The Wellness Motivation Intervention Promoting Physical Activity & Heart Health in Older Latinas. Research in Gerontological Nursing. Accepted.
- [Background] Perez A, Fleury J. Using a Cultural Framework to Assess Motivation for Physical Activity Among Older Hispanic Women: Application of the PEN-3 Model. Fam Community Health. 2018 Jan/Mar;41(1):10-17. doi: 10.1097/FCH.0000000000000176. PMID 29135790
- [Background] Perez A, Fleury J. Wellness motivation theory in practice. Geriatr Nurs. 2009 Mar-Apr;30(2 Suppl):15-20. doi: 10.1016/j.gerinurse.2009.02.006. No abstract available. PMID 19345859
- [Background] Perez A. Culturally Adapting a Timed Activity Intervention for Older Latinos with Dementia and Their Caregivers: Focus Group Results. Clinical Nursing Research. In Review.
- [Background] Nielsen L, Riddle M, King JW; NIH Science of Behavior Change Implementation Team; Aklin WM, Chen W, Clark D, Collier E, Czajkowski S, Esposito L, Ferrer R, Green P, Hunter C, Kehl K, King R, Onken L, Simmons JM, Stoeckel L, Stoney C, Tully L, Weber W. The NIH Science of Behavior Change Program: Transforming the science through a focus on mechanisms of change. Behav Res Ther. 2018 Feb;101:3-11. doi: 10.1016/j.brat.2017.07.002. Epub 2017 Jul 6. PMID 29110885
- [Background] Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. Clin Psychol Sci. 2014 Jan 1;2(1):22-34. doi: 10.1177/2167702613497932. PMID 25821658
- [Background] Wu S. Latinos & Alzheimer's Disease.
- [Background] DeCarli C. Mild cognitive impairment: prevalence, prognosis, aetiology, and treatment. Lancet Neurol. 2003 Jan;2(1):15-21. doi: 10.1016/s1474-4422(03)00262-x. PMID 12849297
- [Background] Unverzagt FW, Sujuan Gao, Lane KA, Callahan C, Ogunniyi A, Baiyewu O, Gureje O, Hall KS, Hendrie HC. Mild cognitive dysfunction: an epidemiological perspective with an emphasis on African Americans. J Geriatr Psychiatry Neurol. 2007 Dec;20(4):215-26. doi: 10.1177/0891988707308804. PMID 18004008
- [Background] Morris JC, Storandt M, Miller JP, McKeel DW, Price JL, Rubin EH, Berg L. Mild cognitive impairment represents early-stage Alzheimer disease. Arch Neurol. 2001 Mar;58(3):397-405. doi: 10.1001/archneur.58.3.397. PMID 11255443
- [Background] Petersen RC. Challenges of epidemiological studies of mild cognitive impairment. Alzheimer Dis Assoc Disord. 2004 Jan-Mar;18(1):1-2. doi: 10.1097/00002093-200401000-00001. No abstract available. PMID 15195456
- [Background] O'Bryant SE, Humphreys JD, Schiffer RB, Sutker PB. Presentation of Mexican Americans to a memory disorder clinic. Journal of Psychopathology and Behavioral Assessment. 2007;29(3):137.
- [Background] National Center for Health Statistics (US). Health, United States, 2015: With Special Feature on Racial and Ethnic Health Disparities. Hyattsville (MD): National Center for Health Statistics (US); 2016 May. Report No.: 2016-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK367640/ PMID 27308685
- [Background] Hebert LE, Weuve J, Scherr PA, Evans DA. Alzheimer disease in the United States (2010-2050) estimated using the 2010 census. Neurology. 2013 May 7;80(19):1778-83. doi: 10.1212/WNL.0b013e31828726f5. Epub 2013 Feb 6. PMID 23390181
- [Background] Wu S, Vega W, Resendez J, Jin H. Latinos & Alzheimer's disease: New numbers behind the crisis. Projection of the costs for US Latinos living with Alzheimer's disease through. 2016;2060.
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Nakakubo S, Makizako H, Doi T, Tsutsumimoto K, Lee S, Lee S, Hotta R, Bae S, Suzuki T, Shimada H. Impact of poor sleep quality and physical inactivity on cognitive function in community-dwelling older adults. Geriatr Gerontol Int. 2017 Nov;17(11):1823-1828. doi: 10.1111/ggi.12973. Epub 2017 Feb 11. PMID 28188962
- [Background] Piercy KL, Troiano RP. Physical Activity Guidelines for Americans From the US Department of Health and Human Services. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e005263. doi: 10.1161/CIRCOUTCOMES.118.005263. No abstract available. PMID 30571339
- [Background] Colcombe SJ, Erickson KI, Scalf PE, Kim JS, Prakash R, McAuley E, Elavsky S, Marquez DX, Hu L, Kramer AF. Aerobic exercise training increases brain volume in aging humans. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1166-70. doi: 10.1093/gerona/61.11.1166. PMID 17167157
- [Background] Kramer AF, Erickson KI, Colcombe SJ. Exercise, cognition, and the aging brain. J Appl Physiol (1985). 2006 Oct;101(4):1237-42. doi: 10.1152/japplphysiol.00500.2006. Epub 2006 Jun 15. PMID 16778001
- [Background] Naismith SL, Hickie IB, Terpening Z, Rajaratnam SM, Hodges JR, Bolitho S, Rogers NL, Lewis SJ. Circadian misalignment and sleep disruption in mild cognitive impairment. J Alzheimers Dis. 2014;38(4):857-66. doi: 10.3233/JAD-131217. PMID 24100124
- [Background] Tranah GJ, Blackwell T, Stone KL, Ancoli-Israel S, Paudel ML, Ensrud KE, Cauley JA, Redline S, Hillier TA, Cummings SR, Yaffe K; SOF Research Group. Circadian activity rhythms and risk of incident dementia and mild cognitive impairment in older women. Ann Neurol. 2011 Nov;70(5):722-32. doi: 10.1002/ana.22468. PMID 22162057
- [Background] Buman MP, King AC. Exercise as a treatment to enhance sleep. American Journal of Lifestyle Medicine. 2010;4(6):500-514.
- [Background] Blumenthal JA, Sherwood A, Babyak MA, Watkins LL, Waugh R, Georgiades A, Bacon SL, Hayano J, Coleman RE, Hinderliter A. Effects of exercise and stress management training on markers of cardiovascular risk in patients with ischemic heart disease: a randomized controlled trial. JAMA. 2005 Apr 6;293(13):1626-34. doi: 10.1001/jama.293.13.1626. PMID 15811982
- [Background] Cricco M, Simonsick EM, Foley DJ. The impact of insomnia on cognitive functioning in older adults. J Am Geriatr Soc. 2001 Sep;49(9):1185-9. doi: 10.1046/j.1532-5415.2001.49235.x. PMID 11559377
- [Background] Eaker ED, Pinsky J, Castelli WP. Myocardial infarction and coronary death among women: psychosocial predictors from a 20-year follow-up of women in the Framingham Study. Am J Epidemiol. 1992 Apr 15;135(8):854-64. doi: 10.1093/oxfordjournals.aje.a116381. PMID 1585898
- [Background] Beaulieu-Bonneau S, Hudon C. Sleep disturbances in older adults with mild cognitive impairment. Int Psychogeriatr. 2009 Aug;21(4):654-66. doi: 10.1017/S1041610209009120. Epub 2009 May 11. PMID 19426575
- [Background] Eakin EG, Bull SS, Riley KM, Reeves MM, McLaughlin P, Gutierrez S. Resources for health: a primary-care-based diet and physical activity intervention targeting urban Latinos with multiple chronic conditions. Health Psychol. 2007 Jul;26(4):392-400. doi: 10.1037/0278-6133.26.4.392. PMID 17605558
- [Background] Grassi K, Gonzalez MG, Tello P, He G. La Vida Caminando: a community-based physical activity program designed by and for rural Latino families. Journal of Health Education. 1999;30(sup2):S13-S17.
- [Background] Marquez DX, Bustamante EE, Aguinaga S, Hernandez R. BAILAMOS: Development, Pilot Testing, and Future Directions of a Latin Dance Program for Older Latinos. Health Educ Behav. 2015 Oct;42(5):604-10. doi: 10.1177/1090198114543006. Epub 2014 Aug 9. PMID 25108538
- [Background] Marquez DX, Wilbur J, Hughes SL, Berbaum ML, Wilson RS, Buchner DM, McAuley E. B.A.I.L.A. - a Latin dance randomized controlled trial for older Spanish-speaking Latinos: rationale, design, and methods. Contemp Clin Trials. 2014 Jul;38(2):397-408. doi: 10.1016/j.cct.2014.06.012. Epub 2014 Jun 24. PMID 24969395
- [Background] Ickes MJ, Sharma M. A systematic review of physical activity interventions in Hispanic adults. J Environ Public Health. 2012;2012:156435. doi: 10.1155/2012/156435. Epub 2012 Feb 8. PMID 22496702
- [Background] Perez A, Fleury J, Keller C. Review of intervention studies promoting physical activity in Hispanic women. West J Nurs Res. 2010 Apr;32(3):341-62. doi: 10.1177/0193945909351300. Epub 2009 Dec 29. PMID 20040732
- [Background] van der Bij AK, Laurant MG, Wensing M. Effectiveness of physical activity interventions for older adults: a review. Am J Prev Med. 2002 Feb;22(2):120-33. doi: 10.1016/s0749-3797(01)00413-5. PMID 11818183
- [Background] Robbins LB, Pender NJ, Conn VS, Frenn MD, Neuberger GB, Nies MA, Topp RV, Wilbur J. Physical activity research in nursing. J Nurs Scholarsh. 2001;33(4):315-21. doi: 10.1111/j.1547-5069.2001.00315.x. PMID 11775300
- [Background] Dergance JM, Calmbach WL, Dhanda R, Miles TP, Hazuda HP, Mouton CP. Barriers to and benefits of leisure time physical activity in the elderly: differences across cultures. J Am Geriatr Soc. 2003 Jun;51(6):863-8. doi: 10.1046/j.1365-2389.2003.51271.x. PMID 12757577
- [Background] McAuley E. Self-efficacy and the maintenance of exercise participation in older adults. J Behav Med. 1993 Feb;16(1):103-13. doi: 10.1007/BF00844757. PMID 8433355
- [Background] Juarbe T, Turok XP, Perez-Stable EJ. Perceived benefits and barriers to physical activity among older Latina women. West J Nurs Res. 2002 Dec;24(8):868-86. doi: 10.1177/019394502237699. PMID 12469724
- [Background] Muse T. Motivation and adherence to exercise for older adults. Topics in Geriatric Rehabilitation. 2005;21(2):107-115.
- [Background] Bandura A. Self-efficacy: The exercise of control. Macmillan; 1997.
- [Background] Heckhausen H. Why some time out might benefit achievement motivation research. In van den Bercken, JHL, Bergen, TCM, De Bruyn, EEJ (Eds.). Achievement and task motivation. Lisse-Holland: Swets & Zeitlinger; 1986.
- [Background] Fleury J, Sedikides C. Wellness motivation in cardiac rehabilitation: the role of self-knowledge in cardiovascular risk modification. Res Nurs Health. 2007 Aug;30(4):373-84. doi: 10.1002/nur.20225. PMID 17654518
- [Background] Schwingel A, Linares DE, Galvez P, Adamson B, Aguayo L, Bobitt J, Castaneda Y, Sebastiao E, Marquez DX. Developing a Culturally Sensitive Lifestyle Behavior Change Program for Older Latinas. Qual Health Res. 2015 Dec;25(12):1733-46. doi: 10.1177/1049732314568323. Epub 2015 Jan 16. PMID 25595148
- [Background] Idali Torres M, Marquez DX, Carbone ET, Stacciarini JM, Foster JW. Culturally responsive health promotion in puerto rican communities: a structuralist approach. Health Promot Pract. 2008 Apr;9(2):149-58. doi: 10.1177/1524839907307675. PMID 18340090
- [Background] Hunter JB, de Zapien JG, Papenfuss M, Fernandez ML, Meister J, Giuliano AR. The impact of a promotora on increasing routine chronic disease prevention among women aged 40 and older at the U.S.-Mexico border. Health Educ Behav. 2004 Aug;31(4 Suppl):18S-28S. doi: 10.1177/1090198104266004. PMID 15296689
- [Background] Mathews AE, Laditka SB, Laditka JN, Wilcox S, Corwin SJ, Liu R, Friedman DB, Hunter R, Tseng W, Logsdon RG. Older adults' perceived physical activity enablers and barriers: a multicultural perspective. J Aging Phys Act. 2010 Apr;18(2):119-40. doi: 10.1123/japa.18.2.119. PMID 20440026
- [Background] Kim S, Flaskerud JH, Koniak-Griffin D, Dixon EL. Using community-partnered participatory research to address health disparities in a Latino community. J Prof Nurs. 2005 Jul-Aug;21(4):199-209. doi: 10.1016/j.profnurs.2005.05.005. PMID 16061166
- [Background] Minkler M, Wallerstein N. Improving health through community organization. Community organizing and community building for health. 2005:26-51.
- [Background] Fleury J. Wellness motivation theory: an exploration of theoretical relevance. Nurs Res. 1996 Sep-Oct;45(5):277-83. doi: 10.1097/00006199-199609000-00005. PMID 8831654
- [Background] Fleury J. The Index of Readiness: development and psychometric analysis. J Nurs Meas. 1994 Winter;2(2):143-54. PMID 7780769
- [Background] Perez A, Fleury J, Shearer N. Salud de Corazon: Cultural Resources for Cardiovascular Health among Older Hispanic Women. Hisp Health Care Int. 2012 Jun 1;10(2):93-100. doi: 10.1891/1540-4153.10.2.93. PMID 23024613
- [Background] Fleury J, Thomas T, Ratledge K. Promoting wellness in individuals with coronary heart disease. J Cardiovasc Nurs. 1997 Apr;11(3):26-42. doi: 10.1097/00005082-199704000-00004. PMID 9095452
- [Background] Wang Y, Song M, Yu L, Wang L, An C, Xun S, Zhao X, Gao Y, Wang X. Mild cognitive impairment: vascular risk factors in community elderly in four cities of Hebei Province, China. PLoS One. 2015 May 11;10(5):e0124566. doi: 10.1371/journal.pone.0124566. eCollection 2015. PMID 25962184
- [Background] Verdelho A, Madureira S, Ferro JM, Baezner H, Blahak C, Poggesi A, Hennerici M, Pantoni L, Fazekas F, Scheltens P, Waldemar G, Wallin A, Erkinjuntti T, Inzitari D; LADIS Study. Physical activity prevents progression for cognitive impairment and vascular dementia: results from the LADIS (Leukoaraiosis and Disability) study. Stroke. 2012 Dec;43(12):3331-5. doi: 10.1161/STROKEAHA.112.661793. Epub 2012 Nov 1. PMID 23117721
- [Background] King AC, King DK. Physical activity for an aging population. Public Health Reviews. 2010;32(2):401.
- [Background] Winchester J, Dick MB, Gillen D, Reed B, Miller B, Tinklenberg J, Mungas D, Chui H, Galasko D, Hewett L, Cotman CW. Walking stabilizes cognitive functioning in Alzheimer's disease (AD) across one year. Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):96-103. doi: 10.1016/j.archger.2012.06.016. Epub 2012 Sep 5. PMID 22959822
- [Background] Marquez DX, Wilson R, Aguinaga S, Vasquez P, Fogg L, Yang Z, Wilbur J, Hughes S, Spanbauer C. Regular Latin Dancing and Health Education May Improve Cognition of Late Middle-Aged and Older Latinos. J Aging Phys Act. 2017 Jul;25(3):482-489. doi: 10.1123/japa.2016-0049. Epub 2017 Jun 28. PMID 28095105
- [Background] Aguinaga S, Marquez DX. Feasibility of a Latin Dance Program for Older Latinos With Mild Cognitive Impairment. Am J Alzheimers Dis Other Demen. 2017 Dec;32(8):479-488. doi: 10.1177/1533317517719500. Epub 2017 Jul 6. PMID 28683560
- [Background] Aguinaga S, Marquez DX. Impact of Latin Dance on Physical Activity, Cardiorespiratory Fitness, and Sedentary Behavior Among Latinos Attending an Adult Day Center. J Aging Health. 2019 Mar;31(3):397-414. doi: 10.1177/0898264317733206. Epub 2017 Sep 27. PMID 29254398
- [Background] Fleury J, Keller C, Perez A. Exploring resources for physical activity in Hispanic women, using photo elicitation. Qual Health Res. 2009 May;19(5):677-86. doi: 10.1177/1049732309334471. PMID 19380503
- [Background] Perez A, Garces A, Hunter RH, Marquez DX. An audit of a diverse community for safe routes to age in place: environmental policy implications. J Gerontol Nurs. 2015 Mar;41(3):13-21. doi: 10.3928/00989134-20150205-01. PMID 25710264
- [Background] Perez A. Physical Activity and Sleep in Older Latinos with Mild Cognitive Impairment. Paper presented at: The Gerontological Society of America2018; Boston, MA.
- [Background] Perez A, Hodgson N. Influence of Community on Well-Being in Home Dwelling Multi-ethnic Older Adults with Dementia. American Public Health Association's 2019 Annual Meeting and Expo; 2019; Philadelphia, PA.
- [Background] Koorts H, Eakin E, Estabrooks P, Timperio A, Salmon J, Bauman A. Implementation and scale up of population physical activity interventions for clinical and community settings: the PRACTIS guide. Int J Behav Nutr Phys Act. 2018 Jun 8;15(1):51. doi: 10.1186/s12966-018-0678-0. PMID 29884236
- [Background] Suarez-Morales L, Matthews J, Martino S, Ball SA, Rosa C, Farentinos C, Szapocznik J, Carroll KM. Issues in designing and implementing a Spanish-language multi-site clinical trial. Am J Addict. 2007 May-Jun;16(3):206-15. doi: 10.1080/10550490701375707. PMID 17612825
- [Background] Krogstad JM, Gonzalez-Barrera A. A majority of English-speaking Hispanics in the US are bilingual. Washington, DC: Pew Research Center. 2015.
- [Background] Martinez CR Jr, McClure HH, Eddy JM, Ruth B, Hyers MJ. Recruitment and retention of Latino immigrant families in prevention research. Prev Sci. 2012 Feb;13(1):15-26. doi: 10.1007/s11121-011-0239-0. PMID 21818583
- [Background] Marín G, Marín BV. Research with Hispanic populations. Research with Hispanic populations. Thousand Oaks, CA, US: Sage Publications, Inc:ix, 130-ix, 130.
- [Background] Resnick B, Ory MG, Hora K, et al. The Exercise Assessment and Screening for You (EASY) tool: application in the oldest old population. American Journal of Lifestyle Medicine. 2008;2(5):432-440.
- [Background] Marcus BH, Dubbert PM, Forsyth LH, McKenzie TL, Stone EJ, Dunn AL, Blair SN. Physical activity behavior change: issues in adoption and maintenance. Health Psychol. 2000 Jan;19(1S):32-41. doi: 10.1037/0278-6133.19.suppl1.32. PMID 10709946
- [Background] Gil L, Ruiz de Sanchez C, Gil F, Romero SJ, Pretelt Burgos F. Validation of the Montreal Cognitive Assessment (MoCA) in Spanish as a screening tool for mild cognitive impairment and mild dementia in patients over 65 years old in Bogota, Colombia. Int J Geriatr Psychiatry. 2015 Jun;30(6):655-62. doi: 10.1002/gps.4199. Epub 2014 Oct 16. PMID 25320026
- [Background] Fleury J, Keller C, Perez A, Lee SM. The role of lay health advisors in cardiovascular risk reduction: a review. Am J Community Psychol. 2009 Sep;44(1-2):28-42. doi: 10.1007/s10464-009-9253-9. PMID 19533327
- [Background] Carrasquillo O, Patberg E, Alonzo Y, Li H, Kenya S. Rationale and design of the Miami Healthy Heart Initiative: a randomized controlled study of a community health worker intervention among Latino patients with poorly controlled diabetes. Int J Gen Med. 2014 Feb 27;7:115-26. doi: 10.2147/IJGM.S56250. eCollection 2014. PMID 24600243
- [Background] Keller C, Fleury J, Perez A, Belyea M, Castro FG. Mujeres en accion: design and baseline data. J Community Health. 2011 Oct;36(5):703-14. doi: 10.1007/s10900-011-9363-9. PMID 21298400
- [Background] National Heart L, Institute B. Su Corazón Su Vida: Manual del Promotor y Promotora de Salud. Bethesda, MD: US Department of Health and Human Services, NIH. 2000.
- [Background] Keller C, Fleury J. Factors related to physical activity in Hispanic women. J Cardiovasc Nurs. 2006 Mar-Apr;21(2):142-5. doi: 10.1097/00005082-200603000-00012. PMID 16601533
- [Background] Lautenschlager NT, Cox KL, Flicker L, Foster JK, van Bockxmeer FM, Xiao J, Greenop KR, Almeida OP. Effect of physical activity on cognitive function in older adults at risk for Alzheimer disease: a randomized trial. JAMA. 2008 Sep 3;300(9):1027-37. doi: 10.1001/jama.300.9.1027. PMID 18768414
- [Background] Office of the Surgeon General (US). Step It Up! The Surgeon General's Call to Action to Promote Walking and Walkable Communities [Internet]. Washington (DC): US Department of Health and Human Services; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK538433/ PMID 30860691
- [Background] Kreuter MW, Skinner CS. Tailoring: what's in a name? Health Educ Res. 2000 Feb;15(1):1-4. doi: 10.1093/her/15.1.1. No abstract available. PMID 10788196
- [Background] Karvonen method.
- [Background] Hunter R, Ivey S, Satariano W, Bayles C. Engaging Older Adults to Be More Active Where They Live: Audit Tool Development.
- [Background] Baker PR, Francis DP, Soares J, Weightman AL, Foster C. Community wide interventions for increasing physical activity. Sao Paulo Medical Journal. 2011;129(6):436-437.
- [Background] Baker PR, Francis DP, Soares J, Weightman AL, Foster C. Community wide interventions for increasing physical activity. Cochrane Database Syst Rev. 2015 Jan 5;1(1):CD008366. doi: 10.1002/14651858.CD008366.pub3. PMID 25556970
- [Background] Wallerstein N, Bernstein E. Empowerment education: Freire's ideas adapted to health education. Health Educ Q. 1988 Winter;15(4):379-94. doi: 10.1177/109019818801500402. PMID 3230016
- [Background] Wallerstein N, Duran B. Community-based participatory research contributions to intervention research: the intersection of science and practice to improve health equity. Am J Public Health. 2010 Apr 1;100 Suppl 1(Suppl 1):S40-6. doi: 10.2105/AJPH.2009.184036. Epub 2010 Feb 10. PMID 20147663
- [Background] Lachman ME, Lipsitz L, Lubben J, Castaneda-Sceppa C, Jette AM. When Adults Don't Exercise: Behavioral Strategies to Increase Physical Activity in Sedentary Middle-Aged and Older Adults. Innov Aging. 2018 Jan;2(1):igy007. doi: 10.1093/geroni/igy007. Epub 2018 Apr 5. PMID 30003146
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Kelly LA, McMillan DG, Anderson A, Fippinger M, Fillerup G, Rider J. Validity of actigraphs uniaxial and triaxial accelerometers for assessment of physical activity in adults in laboratory conditions. BMC Med Phys. 2013 Nov 26;13(1):5. doi: 10.1186/1756-6649-13-5. PMID 24279826
- [Background] Buchman AS, Boyle PA, Yu L, Shah RC, Wilson RS, Bennett DA. Total daily physical activity and the risk of AD and cognitive decline in older adults. Neurology. 2012 Apr 24;78(17):1323-9. doi: 10.1212/WNL.0b013e3182535d35. Epub 2012 Apr 18. PMID 22517108
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] Lee IM, Shiroma EJ. Using accelerometers to measure physical activity in large-scale epidemiological studies: issues and challenges. Br J Sports Med. 2014 Feb;48(3):197-201. doi: 10.1136/bjsports-2013-093154. Epub 2013 Dec 2. PMID 24297837
- [Background] Buchman AS, Wilson RS, Bennett DA. Total daily activity is associated with cognition in older persons. Am J Geriatr Psychiatry. 2008 Aug;16(8):697-701. doi: 10.1097/JGP.0b013e31817945f6. PMID 18669949
- [Background] Miller NE, Strath SJ, Swartz AM, Cashin SE. Estimating absolute and relative physical activity intensity across age via accelerometry in adults. J Aging Phys Act. 2010 Apr;18(2):158-70. doi: 10.1123/japa.18.2.158. PMID 20440028
- [Background] Sallis JF, Johnson MF, Calfas KJ, Caparosa S, Nichols JF. Assessing perceived physical environmental variables that may influence physical activity. Res Q Exerc Sport. 1997 Dec;68(4):345-51. doi: 10.1080/02701367.1997.10608015. PMID 9421846
- [Background] Monsell SE, Dodge HH, Zhou XH, Bu Y, Besser LM, Mock C, Hawes SE, Kukull WA, Weintraub S; Neuropsychology Work Group Advisory to the Clinical Task Force. Results From the NACC Uniform Data Set Neuropsychological Battery Crosswalk Study. Alzheimer Dis Assoc Disord. 2016 Apr-Jun;30(2):134-9. doi: 10.1097/WAD.0000000000000111. PMID 26485498
- [Background] Weintraub S, Salmon D, Mercaldo N, Ferris S, Graff-Radford NR, Chui H, Cummings J, DeCarli C, Foster NL, Galasko D, Peskind E, Dietrich W, Beekly DL, Kukull WA, Morris JC. The Alzheimer's Disease Centers' Uniform Data Set (UDS): the neuropsychologic test battery. Alzheimer Dis Assoc Disord. 2009 Apr-Jun;23(2):91-101. doi: 10.1097/WAD.0b013e318191c7dd. PMID 19474567
- [Background] Randolph C, Tierney MC, Mohr E, Chase TN. The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS): preliminary clinical validity. J Clin Exp Neuropsychol. 1998 Jun;20(3):310-9. doi: 10.1076/jcen.20.3.310.823. PMID 9845158
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Lambiase MJ, Gabriel KP, Chang YF, Kuller LH, Matthews KA. Utility of actiwatch sleep monitor to assess waking movement behavior in older women. Med Sci Sports Exerc. 2014 Dec;46(12):2301-7. doi: 10.1249/MSS.0000000000000361. PMID 24781894
- [Background] Cross S, Markus H. Possible selves across the life span. Human development. 1991;34(4):230-255.
- [Background] Fleury J, Sedikides C, Donovan KD. Possible health selves of older African Americans: Toward increasing the effectiveness of health promotion efforts. Topics in Geriatric Rehabilitation. 2002;18(1):52-58.
- [Background] McMahon SK, Wyman JF, Belyea MJ, Shearer N, Hekler EB, Fleury J. Combining Motivational and Physical Intervention Components to Promote Fall-Reducing Physical Activity Among Community-Dwelling Older Adults: A Feasibility Study. Am J Health Promot. 2016 Nov;30(8):638-644. doi: 10.4278/ajhp.130522-ARB-265. Epub 2016 Jun 16. PMID 26389979
- [Background] Silva-Smith AL, Fleury J, Belyea M. Effects of a physical activity and healthy eating intervention to reduce stroke risk factors in older adults. Prev Med. 2013 Nov;57(5):708-11. doi: 10.1016/j.ypmed.2013.07.004. Epub 2013 Jul 13. PMID 23859934
- [Background] Fleury J. The index of self-regulation: development and psychometric analysis. J Nurs Meas. 1998 Summer;6(1):3-17. PMID 9769608
- [Background] Roy A, Bhaumik DK, Aryal S, Gibbons RD. Sample size determination for hierarchical longitudinal designs with differential attrition rates. Biometrics. 2007 Sep;63(3):699-707. doi: 10.1111/j.1541-0420.2007.00769.x. PMID 17825003
- [Background] Benjamini Y, Drai D, Elmer G, Kafkafi N, Golani I. Controlling the false discovery rate in behavior genetics research. Behav Brain Res. 2001 Nov 1;125(1-2):279-84. doi: 10.1016/s0166-4328(01)00297-2. PMID 11682119
- [Background] Akaike H. A new look at statistical model identification. IEEE Transactions on Automatic Control. 1974;19:716-723.
- [Background] Selig JP, Preacher KJ. Mediation models for longitudinal data in developmental research. Research in Human Development. 2009;6(2-3):144-164.
- [Background] Cheong J, Mackinnon DP, Khoo ST. Investigation of Mediational Processes Using Parallel Process Latent Growth Curve Modeling. Struct Equ Modeling. 2003 Apr 1;10(2):238. doi: 10.1207/S15328007SEM1002_5. PMID 20157639
- [Background] Office of the Inspector General. Medicaid Drug Price Comparison: Average Sales Price To Average Wholesale Price, . Department of Health & Human Services (DHHS); 2005.
- [Background] Gold M, Siegel J, Russell L, Weinstein M, eds. Cost-effectiveness in health and medicine. New York, NY: Oxford University Press; 1996.
- [Background] Glick HA, McElligott S, Pauly MV, Willke RJ, Bergquist H, Doshi J, Fleisher LA, Kinosian B, Perfetto E, Polsky DE, Schwartz JS. Comparative effectiveness and cost-effectiveness analyses frequently agree on value. Health Aff (Millwood). 2015 May;34(5):805-11. doi: 10.1377/hlthaff.2014.0552. PMID 25941282
- [Background] Ramsey S, Willke R, Briggs A, Brown R, Buxton M, Chawla A, Cook J, Glick H, Liljas B, Petitti D, Reed S. Good research practices for cost-effectiveness analysis alongside clinical trials: the ISPOR RCT-CEA Task Force report. Value Health. 2005 Sep-Oct;8(5):521-33. doi: 10.1111/j.1524-4733.2005.00045.x. PMID 16176491